CLINICAL TRIAL: NCT03306394
Title: An Open-label Early Access Phase IIIb Study of Trifluridine / Tipiracil (S 95005/TAS-102) in Patients With a Pretreated Metastatic Colorectal Cancer (PRECONNECT)
Brief Title: A Study of Trifluridine/Tipiracil (Also Known as S 95005 or TAS-102) in Patients With a Pretreated Colorectal Cancer That Has Spread (Metastatic).
Acronym: PRECONNECT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Collaborators: ADIR, a Servier Group company (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL3-95005-004; 2016-002311-18 (EudraCT Number)
Record Dates: First submitted 2017-08-02; First posted 2017-10-11 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Metastatic Colorectal Cancer
Keywords: metastatic; colorectal; cancer; trifluridine/tipiracil; early access
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Neoplasms | interventions — Trifluridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- S95005 (Experimental): Film-coated tablet containing 15 mg of trifluridine and 7.065 mg of tipiracil hydrochloride, or 20 mg of trifluridine and 9.42 mg of tipiracil hydrochloride, taken orally twice a day at the dose of 35 mg/m²/dose. The treatment is given until progression of disease, unacceptable toxicity, investigator decision, patient refusal or until market authorization or reimbursement has been granted by the relevant Authority of the country where that patient is treated or until trifluridine / tipiracil is available by a doctor's prescription or can be accessed from another source or Sponsor decision.
  Interventions: Drug: Trifluridine/Tipiracil hydrochloride (S95005)

INTERVENTIONS:
Drug: Trifluridine/Tipiracil hydrochloride (S95005)

SUMMARY:
The purpose of this study is to collect additional safety and efficacy data during treatment with trifluridine / tipiracil in patients with a pretreated metastatic colorectal cancer (mCRC).

Eligible patients may receive an early access to trifluridine / tipiracil through this clinical study until progression of disease, unacceptable toxicity, investigator decision, patient refusal or until market authorization or reimbursement has been granted by the relevant Authority of the country where that patient is treated or until trifluridine / tipiracil is available by a doctor's prescription or can be accessed from another source or Sponsor decision.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female participant aged ≥18 years old.
* Has definitive histologically confirmed adenocarcinoma of the colon or rectum.
* Has metastatic lesion(s).
* Has received at least 2 prior regimens of standard chemotherapies (including fluoropyrimidines, irinotecan, oxaliplatin, an anti-VEGF monoclonal antibody and at least one of the anti-EGFR monoclonal antibodies for RAS wild-type patients) for mCRC and is refractory or intolerant to those chemotherapies or is not candidate for those chemotherapies.
* Has Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 during the screening period.
* Is able to take medications orally (i.e., no feeding tube).
* Has adequate organ function.
* Women of childbearing potential must have been tested negative in a serum pregnancy test within 7 days prior to first day of test drug administration. Female participants of childbearing potential and male participants with partners of childbearing potential must agree to use a highly effective method of birth control during the study and for 6 months after the discontinuation of study medication. Women and female partners using hormonal contraceptive must also use a barrier method.

Exclusion Criteria:

* Pregnancy, breastfeeding or possibility of becoming pregnant during the study.
* Eligible for enrolment into another available ongoing clinical study of trifluridine / tipiracil.
* Has previously received trifluridine / tipiracil or hypersensitivity to the active substances or to any of the excipients of trifluridine / tipiracil.
* Has rare hereditary problems of galactose intolerance, the Lapp lactase deficiency, or glucose-galactose malabsorption.
* Has certain serious illness or medical condition(s) described in the protocol.
* Has had certain other recent treatment e.g. major surgery, anticancer therapy, radiation therapy, participation in another interventional study, within the specified time frames prior to first day of study drug administration.
* Has unresolved toxicity of greater than or equal to Common Terminology Criteria for Adverse Events (CTCAE) Grade 2 attributed to any prior therapies (excluding anemia, alopecia, skin pigmentation, and platinum-induced neurotoxicity).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 907 (Actual)
Dates: Start 2016-10-18 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events [safety and tolerability] | Through 28 days following last administration of study medication
Abnormalities in laboratory assessment | Through study completion, an average of 12 weeks
Abnormalities in performance status (ECOG) | Through study completion, an average of 12 weeks
Abnormalities in vital signs | Through study completion, an average of 12 weeks

SECONDARY OUTCOMES:
Progression free survival (PFS) | Through study completion, an average of 12 weeks
  time from the date of first study drug intake until the date of the investigator-assessed disease progression or death due to any cause whichever occurs first.
Quality of life using the questionnaire EQ-5D | Through study completion, an average of 12 weeks
Quality of life using the questionnaire EORTC QLQ-C30 | Through study completion, an average of 12 weeks

CONTACTS AND LOCATIONS:
Locations (99):
- Australia (8):
  - Chris O'Brien Lifehouse Oncology, Camperdown
  - St Vincent's Hospital The Kinghorn Cancer Centre, Darlinghurst
  - St Vincent's Hospital (Melbourne) Cancer Centre, Fitzroy
  - The Canberra Hospital Cancer,Ambulatory & Community Health Service (CACHS) Bldg 19, Garran
  - Royal Brisbane & Women's Hospital Clinical Research Unit, Herston
  - Cabrini Hospital Cabrini Haematology and Oncology Centre, Malvern
  - Perth Oncology - Mount Hospital, Perth
  - The Queen Elizabeth Hospital Haematology and Oncology Unit, Woodville
- Belgium (5):
  - Hôpital Universitaire Erasme Gastro-Entérologie, Brussels
  - Cliniques Universitaires St. Luc Oncologie médicale, Brussels
  - Universitair Ziekenhuis Antwerpen Oncologie, Edegem
  - U.Z. Gent Digestieve Oncologie, Ghent
  - UZ Leuven Campus Gasthuisberg Digestieve Oncologie, Leuven
- Brazil (6):
  - Hospital Mãe de Deus Centro Intergrado de Pesquisa, Porto Alegre
  - Clinicas Oncológicas Integradas (COI), Rio de Janeiro
  - AMO Assistencia Multidisciplinar em Oncologia GEM Assistencia Medica Especializada, Salvador
  - Instituto do Cancer do Estado de Sao Paulo - ICESP Núcleo de Pesquisa, São Paulo
  - Hospital A C Camargo Unidade de Pesquisa Clínica, São Paulo
  - Instituto Brasileiro de Controle do Câncer Unidadde de Pesquisa Clínica, São Paulo
- Bulgaria (4):
  - Complex oncology center - Plovdiv, Plovdiv
  - Military Medical Academy - MHAT Oncology clinic, Sofia
  - Specialized hospital for active treatment in oncology, Sofia
  - SHAT of oncology diseases, Varna
- Croatia (2):
  - Klinicki bolnicki centar Rijeka Klinika za radioterapiju i onkologiju, Rijeka
  - Klinicki bolnicki centar Zagreb Klinika za onkologiju, Zagreb
- France (23):
  - Hopital Privé Les Bonnettes Pharmacie centrale, Arras
  - Institut Sainte Catherine Institut Sainte Catherine, Avignon
  - Centre de lutte contre le cancer Francois Baclesse UCP Digestif, Caen
  - Hôpital Trousseau Hépato-gastroentérologie et cancérologie digestive, Chambray-lès-Tours
  - CHU Hôpital du Bocage/ François Mitterrand Hépato-gastroentérologie, Dijon
  - CHU de Grenoble Oncologie médicale Hépato-gastroentérologie - 7D, Grenoble
  - CHD - Les Oudairies service d'hepato-gastroenterologie, La Roche-sur-Yon
  - Franco-British Institue Department of Medical Oncology, Levallois-Perret
  - Hopital Privé Jean Mermoz Service de Gastro entérologie et d'Oncologie médicale, Lyon
  - CRLCC Léon Bérard Service d'Oncologie, Lyon
  - CHU de la Timone Hépato-Gastro-Entérologie, Marseille
  - Hôpital Nord Franche-Comté - Site du Mittan Service d'oncologie médicale, Montbéliard
  - CRLCC Val d'Aurelle Oncologie Médicale, Montpellier
  - Centre Antoine Lacassagne Dpt d'Oncologie Médicale, Nice
  - Hôpital Saint-Antoine Service d'Oncologie Médicale, Paris
  - Hôpital Européen Georges Pompidou Oncologie Hépatogastroenterologie-oncologie digestive, Paris
  - Groupe Hospitalier Pitié Salpêtrière Service d'hépato-gastro-entérologie, Paris
  - Hôpital Haut-Lévèque Hépato-gastroentérologie et oncologie digestive, Pessac
  - CHU de Poitiers Pole Régional de Cancérologie, Poitiers
  - CHU Robert DEBRE service d'hepato-gastroenterologie / Cancérologie Digestive, Reims
  - Centre Eugène Marquis Service d'Oncologie Médicale, Rennes
  - Hôpital Nord Pôle Digestif Urologie-Andrologie, Saint-Etienne
  - CHU Toulouse Rangueil Oncologie médicale digestive, Toulouse
- Ireland (2):
  - Bon Secours Hospital, Cork
  - The Adelaide and Meath Hospital, Dublin
- Italy (18):
  - Ist.Tumori "Giovanni Paolo II" IRCCS Osp.Oncologico di Bari U.O.C. di Oncologia Medica, Bari
  - Fondazione Poliambulanza Istituto Ospedaliero Clinical Oncology, Brescia
  - ARNAS - Azienda Ospedaliera Garibaldi - Nesima Struttura Complessa di Oncologia Medica, Catania
  - Azienda Ospedaliero-Universitaria Careggi Struttura Complessa Oncologia Medica, Florence
  - Ist.Scientifico Romagnolo per lo Studio e la Cura dei Tumori Department of Clinical Oncology, Meldola
  - Fondazione IRCCS Istituto Nazionale dei Tumori S.S. Oncologia Medica Gastrenterologia, Milan
  - A.O.U. Seconda Università degli Studi di Napoli U.O.C. di Oncologia Medica e di Ematologia, Napoli
  - Istituto Oncologico Veneto IOV - IRCCS Unità Operativa Complessa Oncologia Medica 1, Padua
  - Azienda Ospedaliera "Civico-Di Cristina" - Ospedale Civico Oncologia Medica, Palermo
  - Ospedale Civile Santo Spirito Struttura Complessa di Oncologia Medica, Pescara
  - A.O.U. Pisana-Ospedale Santa Chiara U.O. di Oncologia Medica 2, Pisa
  - Arcispedale Santa Maria Nuova Unità di Oncologia, Reggio Emilia
  - Ospedale INFERMI Reparto di Oncologia, Rimini
  - Policlinico Universitario Campus Biomedico UOC di Oncologia Medica, Roma
  - Policlinico Universitario Agostino Gemelli U.O.C. di Oncologia Medica, Roma
  - Istituto Clinico Humanitas I.R.C.C.S Dipartimento di Oncologia Medica ed Ematologia, Rozzano (MI)
  - IRCSS Casa Sollievo della Sofferenza Dipartimento Onco-Ematologia, San Giovanni Rotondo
  - A.O.U. Città della Salute e della Scienza di Torino S.C. Oncologia Medica 1 - Colo-Rectal Cancer Unit, Torino
- Centro Hemato-Oncologico de Panama, Panama City, Panama
- Poland (6):
  - Bialostockie Centrum Onkologii im Marii Curie-Sklodowskiej Oddzial Onkologii Klinicznej im Dr Ewy Pileckiej z pododdzialem Chemioterapii Dziennej, Bialystok
  - Uniwersyteckie Centrum Kliniczne Klinika Onkologii i Radioterapii, Gdansk
  - Opolskie Centrum Onkologii im. Tadeusza Koszarowskiego Oddzial Onkologii Klinicznej, Opole
  - Wielkopolskie Centrum Onkologii im Marii Sklodowskiej-Curie Oddzial Chemioterapii, Poznan
  - Centrum Onkologii - Instytut im. Marii Sklodowskiej-Curie Klinika Gastroenterologii Onkologicznej, Warsaw
  - Magodent Sp. z o.o., Warsaw
- Portugal (6):
  - Hospital Garcia de Orta Serviço de Oncologia Médica, Almada
  - Centro Hospitalar e Universitário de Comibra E.P.E. Serviço de Oncologia Médica, Coimbra
  - Instituto Português de Oncologia de Coimbra Serviço de Oncologia Médica, Coimbra
  - Centro Hospitalar de Lisboa Norte E.P.E. - H. Santa Maria Serviço de Oncologia Médica, Lisbon
  - Instituto Português de Oncologia do Porto Serviço de Oncologia Médica, Porto
  - Centro Hospitalar de São João E.P.E. Serviço de Oncologia, Porto
- Romania (3):
  - Spitalul Clinic "Fundeni" Departament Oncologie Medicala - Gastroenterologie, Bucharest
  - Institutul Oncologic "Prof. Dr. I. Chiricuta" Cluj Napoca Oncologie Medicala, Cluj-Napoca
  - Institutul Regional de Oncologie Iasi Clinica de Oncologie Medicala, Iași
- Slovakia (2):
  - Onkologicky ustav sv. Alzbety,s.r.o. Interna Klinika VSZ a SP a OUSA, Bratislava
  - Vychodoslovensky onkologicky ustav Oddelenie klinickej onkologie, Košice
- Onkoloski Institut Ljubljana, Ljubljana, Slovenia
- Turkey (Türkiye) (8):
  - Gazi University Faculty of Medicine Medical Oncology Department, Ankara
  - Hacettepe University Faculty of Medicine, Ankara
  - Uludag University Faculty of Medicine, Bursa
  - Trakya University Faculty of Medicine, Edirne
  - Istanbul University, Istanbul
  - Marmara University Pendik Training and Research Hospital, Istanbul
  - Ege University Faculty of Medicine Medical Oncology Department, Izmir
  - Erciyes University Mehmet Kemal Dedeman Hematology Oncology, Kayseri
- Ukraine (4):
  - Kharkiv Regional Oncology Center, Kharkiv
  - Kyiv City Clinical Oncological Centre Day care facility, Kiev
  - Clinical and diagn.Centre of Medics-rey Inter. Group LLC - Hospital of Israeli Oncology "LISOD, Kyiv
  - Treatment-diagnostic Centre PJSC "House of medicine", Odesa

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: http://clinicaltrials.servier.com

REFERENCES:
- [Background] Bachet JB, Wyrwicz L, Price T, Cremolini C, Phelip JM, Portales F, Ozet A, Cicin I, Atlan D, Becquart M, Vidot L, Mounedji N, Van Cutsem E, Taieb J, Falcone A. Safety, efficacy and patient-reported outcomes with trifluridine/tipiracil in pretreated metastatic colorectal cancer: results of the PRECONNECT study. ESMO Open. 2020 Jun;5(3):e000698. doi: 10.1136/esmoopen-2020-000698. PMID 32487542
- [Derived] Taieb J, Price T, Vidot L, Chevallier B, Wyrwicz L, Bachet JB. Safety and efficacy of trifluridine/tipiracil in previously treated metastatic colorectal cancer: final results from the phase IIIb single-arm PRECONNECT study by duration of therapy. BMC Cancer. 2023 Jan 27;23(1):94. doi: 10.1186/s12885-022-10489-4. PMID 36707808
- [Derived] Ozet A, Dane F, Aykan NF, Yalcin S, Evrensel T, Ozkan M, Karabulut B, Ormeci MN, Atasev O, Vidot L, Cicin I. Safety and efficacy of trifluridine/tipiracil in previously treated metastatic colorectal cancer: PRECONNECT Turkey. Future Oncol. 2022 Sep;18(29):3267-3276. doi: 10.2217/fon-2022-0455. Epub 2022 Aug 30. PMID 36040321
- [Derived] Zaniboni A, Barone CA, Banzi MC, Bergamo F, Blasi L, Bordonaro R, Bartolomeo MD, Costanzo FD, Frassineti GL, Garufi C, Giuliani F, Latiano TP, Martinelli E, Personeni N, Racca P, Tamburini E, Tonini G, Besse MG, Spione M, Falcone A. Italian results of the PRECONNECT study: safety and efficacy of trifluridine/tipiracil in metastatic colorectal cancer. Future Oncol. 2021 Jun;17(18):2315-2324. doi: 10.2217/fon-2020-1278. Epub 2021 Mar 5. PMID 33663264
- Available data/document: Individual Participant Data Set — https://clinicaltrials.servier.com/
- Available data/document: Study Protocol — https://clinicaltrials.servier.com/
- Available data/document: Statistical Analysis Plan — https://clinicaltrials.servier.com/
- Available data/document: Informed Consent Form — https://clinicaltrials.servier.com/
- Available data/document: Clinical Study Report — https://clinicaltrials.servier.com/
- Available data/document: study-level clinical trial data — https://clinicaltrials.servier.com/